CLINICAL TRIAL: NCT07013032
Title: Diagnostic and Prognostic Value of Reticulated Platelet Fraction in Patients With Ventilator-Associated Pneumonia: A Prospective Observational Study
Brief Title: Diagnostic and Prognostic Value of Reticulated Platelet Fraction in Ventilator-Associated Pneumonia (REPLAY-VAP)
Acronym: REPLAY-VAP
Status: Recruiting | Type: Observational
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, HASAN ŞENAY, Dr. Hasan Şenay, Principal Investigator, Department of Intensive Care Medicine, Konya City Hospital TURKEY, Konya City Hospital
Other Study IDs: KSH-RP-VAP-2025-01
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Ventilator-Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ventilator-associated pneumonia (VAP) is a serious infection that occurs in patients who have been on mechanical ventilation for more than 48 hours in the intensive care unit (ICU). Early and accurate diagnosis is critical to reduce complications and improve outcomes. This prospective observational study aims to evaluate the diagnostic and prognostic value of reticulated platelet fraction (RP%) in patients diagnosed with VAP. Blood samples will be taken as part of routine care, and RP% levels will be analyzed using a standard hematology analyzer. The study will investigate whether RP% can help identify VAP earlier and predict outcomes such as mortality and response to antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Receiving mechanical ventilation for more than 48 hours
* Diagnosed with ventilator-associated pneumonia (VAP) according to clinical, radiologic, and laboratory criteria

Exclusion Criteria:

* Diagnosis of pneumonia upon ICU admission
* Pneumonia as the primary reason for initiation of mechanical ventilation
* Mechanical ventilation duration less than 48 hours
* Pregnant or breastfeeding patients
* Presence of chronic inflammatory conditions, hematologic disorders, malignancy, autoimmune disease, or immunosuppressive/chemotherapy/radiotherapy treatment within the past 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adult patients (aged 18 years and older) who are mechanically ventilated for more than 48 hours in the intensive care unit and diagnosed with ventilator-associated pneumonia (VAP).
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of reticulated platelet fraction (RP%) in diagnosing ventilator-associated pneumonia (VAP) | Within 48 hours of VAP diagnosis
  Diagnostic performance of reticulated platelet fraction (RP%) measured as percentage (%) using the Sysmex XN-1000 hematology analyzer (from EDTA-anticoagulated whole blood). The outcome will be evaluated based on sensitivity, specificity, and area under the receiver operating characteristic curve (AUC) for VAP diagnosis, using established clinical and microbiological criteria as the reference standard.

SECONDARY OUTCOMES:
Correlation between baseline RP% and 28-day all-cause mortality | 28 days from VAP diagnosis
  Correlation between reticulated platelet fraction (RP%) measured by Sysmex XN-1000 hematology analyzer and 28-day all-cause mortality. Mortality will be recorded as a binary outcome (alive or dead at day 28), and correlation will be assessed using Spearman or point-biserial correlation coefficients, as appropriate.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Karatay, Turkey (Türkiye)

DOCUMENTS (1):
  • Study Protocol (2025-06-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT07013032/Prot_000.pdf